CLINICAL TRIAL: NCT00528424
Title: A Phase 3, Open-Label Extension Study of the Safety and Efficacy of AA4500 in the Treatment of Subjects With Advanced Dupuytren's Disease
Brief Title: AA4500 (XIAFLEX™, Proposed Name) in the Treatment of Advanced Dupuytren's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AUX-CC-858
Record Dates: First submitted 2007-09-11; First posted 2007-09-12 (Estimated); Results first posted 2010-10-22 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-10

CONDITIONS: Advanced Dupuytren's Disease
MeSH Terms: interventions — Microbial Collagenase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AA4500 0.58 mg (Experimental)
  Interventions: Biological: AA4500

INTERVENTIONS:
Biological: AA4500 — Subjects may have received up to five injections of AA4500 0.58 mg into the cords of the affected hand, with each injection separated by at least 30 days. Individual cords may have received up to a maximum of three AA4500 injections.
  Other Names: XIAFLEX®

SUMMARY:
Study AUX-CC-858 was an open-label continuation of the double-blind Study AUX-CC-857 (NCT00528606). Subjects who complete the Day 90 visit after their initial injection in Study AUX-CC-857 (NCT00528606) entered into Study AUX-CC-858. Subjects who required further treatment in Study AUX-CC-858, either because their treated metacarpophalangeal and/or proximal interphalangeal (PIP) joints did not have a reduction in contracture to 5° or less, the cord affecting that joint received less than three injections of AA4500, or they had other eligible cords that received no treatment in AUX-CC-857 (NCT00528606), had the option to receive up to five injections of AA4500 in this extension study. Subjects requiring further treatment were followed for efficacy and safety on Days 1, 7, and 30 after each injection, with injections separated by four weeks. Follow-up visits for the determination of efficacy and safety were conducted on Day 90, Month 6, and Month 9.

This study was designed to be part of the larger clinical program, for adult patients with Dupuytren's contracture with a palpable cord, where the data from 2 pivotal Placebo-Controlled studies (AUX-CC-857 (NCT00528606) and AUX-CC-859 (NCT00533273)) and 7 non-pivotal studies were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of advanced Dupuytren's disease, with a fixed flexion deformity of at least one finger, other than the thumb, that had a contracture at least 20°, but not greater than 100° for MP (80° for PIP) joints, caused by a palpable cord.
* Had a positive "table top test," defined as the inability to simultaneously place the affected finger(s) and palm flat against a table top.
* Were naïve to AA4500 treatment or had received only one or two injections of AA4500 for the treatment of advanced Dupuytren's disease in AUX-CC-857 ((NCT00528606).
* Were judged to be in good health.
* Must have participated in protocol AUX-CC-857 (NCT00528606).

Exclusion Criteria:

* Had a chronic muscular, neurological, or neuromuscular disorder that affected the hands.
* Had received treatment for advanced Dupuytren's disease within 90 days of enrollment on the joint selected for the initial injection of AA4500, including surgery (fasciectomy or surgical fasciotomy), needle aponeurotomy/fasciotomy, or injection of verapamil and/or interferon.
* Had a known recent history of stroke, bleeding, a disease process that affected the hands, or other medical condition, which in the investigator's opinion, would make the subject unsuitable for enrollment in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2007-12 (Actual); Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Urdaneta, MD, Study Director — Endo Pharmaceuticals
Locations (15):
- United States (15):
  - 100 UCLA Medical Plaza, Suite 305, Los Angeles, California
  - Hand Surgery Clinic, Palo Alto, California
  - Hand Surgery Associates, PC, Denver, Colorado
  - The Hand and Upper Extremity Center of Georgia, P.C., Atlanta, Georgia
  - Rockford Orthopedic Associates, Ltd., Rockford, Illinois
  - The Indiana Hand Center, Indianapolis, Indiana
  - Brigham and Women's Hospital, Department of Orthopedic Surgery, Boston, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - TRIA Orthopaedic Center, Minneapolis, Minnesota
  - Hospital for Special Surgery, New York, New York
  - SUNY Stony Brook - Department of Orthopedics, Stony Brook, New York
  - Health Research Institute, Oklahoma City, Oklahoma
  - Hand Microsurgery & Reconstructive Orthopaedics, Erie, Pennsylvania
  - University Orthopedics Center, State College, Pennsylvania
  - Department of Orthopaedics, Brown University, Rhode Island Hospital, Providence, Rhode Island

REFERENCES:
- See also: XIAFLEX Prescribing Information — http://www.accessdata.fda.gov/drugsatfda_docs/label/2010/125338lbl.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- AA4500 0.58 mg: Collagenase clostridium histolyticum 0.58 mg injected into metacarpophalangeal (MP) and/or proximal interphalangeal (PIP) joints
Period: Overall Study
Arm/Group | AA4500 0.58 mg
Started | 286
Completed | 257
Not Completed | 29
Not completed — Lost to Follow-up | 13
Not completed — Withdrew consent | 2
Not completed — Administrative reason | 2
Not completed — Other | 12

BASELINE CHARACTERISTICS:
Groups:
- AA4500 0.58 mg: Collagenase clostridium histolyticum 0.58 mg injected into MP and/or PIP joints
Arm/Group | AA4500 0.58 mg
Number analyzed (Participants) | 286
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 166
  >=65 years | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 226
Race/Ethnicity, Customized [Number; unit: participants]
  White | 285
  Hispanic | 1
Region of Enrollment [Number; unit: participants]
  United States | 286

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Contracture to 5° or Less
Description: Successfully treated or clinical success in non-primary joints defined as reduction in contracture to within 0-5° of normal within 30 days of injection.
Time Frame: Within 30 days after last injection
Population: Evaluable non-primary joints treated with AA4500 with baseline fixed flexion contracture >5° and at least 1 post-injection contracture measurement. For the purpose of analysis, 13 subjects with non-primary joints treated with AA4500 in double-blind study AUX-CC-857 are included in overall number of participants.
Measure: Number; unit: Percentage of joints
Units Other Than Participants: Joints
Arm/Group | AA4500 0.58 mg
Number analyzed (Participants) | 299
Number analyzed (Joints) | 320
Percentage of joints | 41.9

2. Secondary Outcome: Clinical Improvement After the Last Injection
Description: Clinical improvement in non-primary joints defined as ≥50% reduction from baseline in the degree of contracture within 30 days after injection
Time Frame: Baseline, within 30 days after last injection
Population: as for outcome 1
Measure: Number; unit: Percentage of joints
Units Other Than Participants: Joints
Arm/Group | AA4500 0.58 mg
Number analyzed (Participants) | 299
Number analyzed (Joints) | 320
Percentage of joints | 65.0

3. Secondary Outcome: Percent Reduction From Baseline Contracture After the Last Injection
Description: Percent change in degree of contracture in non-primary joints measured as 100 * (baseline contracture - last available post-injection contracture)/baseline contracture.
Time Frame: Baseline, Day 30 after last injection
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of change
Units Other Than Participants: Joints
Arm/Group | AA4500 0.58 mg
Number analyzed (Participants) | 299
Number analyzed (Joints) | 320
Percentage of change | 60.8 (39.00)

4. Secondary Outcome: Change From Baseline Range of Motion After the Last Injection
Description: Change in degree of range of motion in non-primary joints measured as last available post-injection range of motion - baseline range of motion
Time Frame: Baseline, Day 30 after last injection
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Degrees
Units Other Than Participants: Joints
Arm/Group | AA4500 0.58 mg
Number analyzed (Participants) | 299
Number analyzed (Joints) | 320
Degrees | 24.0 (20.83)

5. Secondary Outcome: Time to Reach Clinical Success
Description: Clinical success in non-primary joints defined as reduction in contracture to within 0-5° of normal within 30 days of injection, displayed in post injection time point categories
Time Frame: Within 30 days after last injection
Population: as for outcome 1
Measure: Number; unit: Percentage of Joints
Units Other Than Participants: Joints
Arm/Group | AA4500 0.58 mg
Number analyzed (Participants) | 299
Number analyzed (Joints) | 320
Percentage of Joints
  Injection 1, Day 1 | 12.5
  Injection 1, Day 7 | 15.9
  Injection 1, Day 30 | 5.9
  Injection 2, Day 0 | 0.0
  Injection 2, Day 1 | 2.2
  Injection 2, Day 7 | 1.3
  Injection 2, Day 30 | 1.9
  Injection 3, Day 0 | 0.0
  Injection 3, Day 1 | 1.3
  Injection 3, Day 7 | 0.6
  Injection 3, Day 30 | 0.3
  Did not reach Clinical Success | 58.1

6. Secondary Outcome: Clinical Success After the First Injection
Description: Clinical success in non-primary joints defined as reduction in contracture to within 0-5° of normal within 30 days of injection.
Time Frame: Within 30 days after first injection
Population: as for outcome 1
Measure: Number; unit: Percentage of Joints
Units Other Than Participants: Joints
Arm/Group | AA4500 0.58 mg
Number analyzed (Participants) | 299
Number analyzed (Joints) | 320
Percentage of Joints | 34.1

7. Secondary Outcome: Clinical Improvement After the First Injection
Description: as for outcome 2
Time Frame: Baseline, within 30 days after first injection
Population: as for outcome 1
Measure: Number; unit: Percentage of Joints
Units Other Than Participants: Joints
Arm/Group | AA4500 0.58 mg
Number analyzed (Participants) | 299
Number analyzed (Joints) | 320
Percentage of Joints | 56.3

8. Secondary Outcome: Percent Reduction From Baseline Contracture After the First Injection
Description: as for outcome 3
Time Frame: Baseline, Day 30 after first injection
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of change
Units Other Than Participants: Joints
Arm/Group | AA4500 0.58 mg
Number analyzed (Participants) | 299
Number analyzed (Joints) | 320
Percentage of change | 53.9 (38.64)

9. Secondary Outcome: Change From Baseline Range of Motion After the First Injection
Description: as for outcome 4
Time Frame: Baseline, Day 30 after first injection
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Degrees
Units Other Than Participants: Joints
Arm/Group | AA4500 0.58 mg
Number analyzed (Participants) | 299
Number analyzed (Joints) | 320
Degrees | 20 (19.46)

ADVERSE EVENTS:
Time Frame: From the time of study drug administration until 30 days after completion of or discharge from the study
Description: This study was designed to be part of the larger clinical program. For information regarding XIAFLEX-associated Serious and Non-serious Adverse events please refer to the XIAFLEX Medication Guide & XIAFLEX Prescribing Information (see links above)
Groups:
- AA4500 0.58 mg: collagenase clostridium histolyticum 0.58mg injected into metacarpophalangeal (MP) and/or proximal interphalangeal (PIP) joints
Arm/Group | AA4500 0.58 mg
Serious Adverse Events (participants affected / at risk) | 9/286
Other Adverse Events (participants affected / at risk) | 171/286
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AA4500 0.58 mg (N=286)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Clostridial infection (Infections and infestations) | 1 (1)
Finger deformity (Musculoskeletal and connective tissue disorders) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Syncope (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AA4500 0.58 mg (N=286)
Blood blister (Skin and subcutaneous tissue disorders) | 21 (22)
Contusion (Injury, poisoning and procedural complications) | 95 (205)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 15 (15)
Ecchymosis (Skin and subcutaneous tissue disorders) | 39 (67)
Injection site haemorrhage (General disorders) | 52 (95)
Injection site pain (General disorders) | 47 (74)
Injection site pruritus (General disorders) | 15 (26)
Injection site swelling (General disorders) | 34 (56)
Oedema peripheral (General disorders) | 136 (386)
Pain (General disorders) | 15 (27)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 66 (98)
Pruritus (Skin and subcutaneous tissue disorders) | 33 (51)
Skin laceration (Injury, poisoning and procedural complications) | 24 (30)
Tenderness (General disorders) | 43 (75)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Auxilium Pharmaceuticals, Inc. agreements may vary with individual investigators but will not prohibit any investigator from publishing. Auxilium supports the publication of results from all centers of a multicenter trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.